CLINICAL TRIAL: NCT05278572
Title: e-SMART/EST Telehealth Intervention to Reduce Depression in Older Women With HIV
Brief Title: e-SMART/EST HIV Telehealth Intervention
Acronym: eSMARTEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13391
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Hiv; Depression
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression | interventions — Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: This clinical trial involves a single treatment arm, consisting of 10 women enrolled in a pilot group. The group will meet weekly for 8 weeks. The intervention consists of cognitive-behavioral stress management/expressive supportive therapy (CBSM+) targeting depression among older women with HIV. The group will be co-facilitated by a Psychologist and a Peer.
Masking Description: N/A: Study only has one arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Experimental): Intervention consists of a psychotherapy trial using cognitive-behavioral stress management/expressive supportive therapy to target depression among HIV-positive older women. Dosage: 8 sessions. Frequency: weekly. Duration: 8 weeks.
  Interventions: Behavioral: Stress Management and Relaxation Training/Expressive Supportive Therapy (SMART/EST)

INTERVENTIONS:
Behavioral: Stress Management and Relaxation Training/Expressive Supportive Therapy (SMART/EST) — Cognitive-behavioral stress management/expressive supportive therapy (CBSM+) group targeting depression

SUMMARY:
The goal of this project is to adapt an evidence-based, enhanced cognitive-behavioral stress management intervention (CSBM+) to target depression among older HIV-positive women in the Bronx, New York. The intervention, "Stress Management and Relaxation Training/Expressive Supportive Therapy" (SMART/EST), demonstrated effectiveness in numerous iterations over 15+ years, including trials with racially diverse HIV-positive women. To meet changing community needs including moving behavioral interventions to telehealth, we will pilot test e-SMART/EST, a teletherapy adaptation with peer support for HIV+ older women.

DETAILED DESCRIPTION:
HIV-positive older women are a neglected, high-risk population for depression. Depression is the most common psychiatric comorbidity for people living with HIV (PLWH), with prevalence between 20-40% and up to 78% in some cohorts. It has associations with lower CD4 (cluster of differentiation 4 - a type of white blood cell) count, higher viral load, reduced medication adherence, and AIDS-related and all-cause mortality. Among older people living with HIV/AIDS (PLWHA), women are more likely than men to be depressed.

Group teletherapy is an efficacious modality to target depression, including among PLWHA, with improved retention and acceptability. To harness these innovations to improve outcomes for HIV+ older women, we will incorporate community feedback to refine and test an online adaption of SMART/EST, an empirically validated cognitive-behavioral stress management/expressive supportive therapy (CBSM+). SMART/EST is effective with HIV+ women and will likely be translated online given the proliferation of cognitive-behavioral therapy (CBT) teletherapy groups. Results will inform secondary prevention with a growing generation of HIV+ older women.

The original, in-person intervention is a 16-session, two-hour weekly group using CBSM+ to target depression, medication adherence, nutrition, physical activity, harm reduction, smoking, and safer sex. e-SMART/EST will be online, condensed to 8 weekly 1-hour sessions, and will target depression. The study has two phases. In Phase 1, we will obtain scientific, community and expert advice from 8 community peer, scientific, and clinical advisors to adapt existent protocols. In Phase 2, we will conduct a pragmatic single group pre-post trial with 10 participants recruited from Montefiore's Women's Interagency HIV Study (WIHS).

e-SMART/EST will be facilitated on MyChart by a Psychologist (PsyD) with prior experience developing the intervention, and co-facilitated by a community peer and Healthy Aging Specialist with 25+ years of experience in HIV programming. Participants will complete pre- and post-test surveys, as well as provide feedback about feasibility, adaptability, and recommendations to improve the intervention. Statistical analyses include paired-samples t-tests and adaptability/feasibility tests, as well as measures of fidelity.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Age 55+
* Teletherapy access
* Depression in last 12 months.
* Fluent in English

Exclusion Criteria:

* HIV-negative or HIV-unknown
* Younger than 55 years old
* Lack of depression in last 12 months
* Non-fluent in English
* Opioid use disorder in last 12 months
* Psychotic disorder in last 12 months.

Ages: 55 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Decrease in score from Baseline in Depression on 21-item Beck Depression Inventory (BDI) at Week 9 | Baseline and Week 9
  The Beck Depression Inventory (BDI) is a validated, self-report 21-item scale assessing depression. Response options range from 0-3 for each item. Item scores are summed, with sum scores ranging from 0-63. Higher scores indicate more depression (i.e., worse outcome). Scale scores from 1-10 indicate: These ups and downs are considered normal; 11-16: Mild mood disturbance; 17-20: Borderline clinical depression; 21-30: Moderate depression; 31-40: Severe depression; over 40: Extreme depression.
Decrease in score from Baseline in Anxiety on 21-item Beck Anxiety Inventory (BAI) at Week 9 | Baseline and Week 9
  The Beck Anxiety Inventory (BAI) is a validated, self-report 21-item scale assessing anxiety. Response options range from 0-3 for each item. Item scores are summed, with sum scores ranging from 0-63. Higher scores indicate more anxiety (i.e., worse outcome). Scale scores from 0-21 indicate: low anxiety; 22-35: moderate anxiety; 36 and above: potentially concerning levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Harris Goldstein, MD, Study Director — Einstein-Rockefeller-City University of New York Center for AIDS Research
Locations (1):
- Albert Einstein College of Medicine - Department of Psychiatry and Behavioral Sciences, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waldron EM, Burnett-Zeigler I, Wee V, Ng YW, Koenig LJ, Pederson AB, Tomaszewski E, Miller ES. Mental Health in Women Living With HIV: The Unique and Unmet Needs. J Int Assoc Provid AIDS Care. 2021 Jan-Dec;20:2325958220985665. doi: 10.1177/2325958220985665. PMID 33472517
- [Result] Jones DL, McPherson-Baker S, Lydston D, Camille J, Brondolo E, Tobin JN, Weiss SM. Efficacy of a group medication adherence intervention among HIV positive women: the SMART/EST Women's Project. AIDS Behav. 2007 Jan;11(1):79-86. doi: 10.1007/s10461-006-9165-8. PMID 17028992
- [Result] Weiss SM, Tobin JN, Antoni M, Ironson G, Ishii M, Vaughn A, Cassells A, Jones D, Schneiderman N, Brondolo E, Laperriere A, Lopez M, Villar-Loubet O, Camille J, Kumar M, Page JB; SMART/EST Women's Project Team*. Enhancing the health of women living with HIV: the SMART/EST Women's Project. Int J Womens Health. 2011 Feb 15;3:63-77. doi: 10.2147/IJWH.S5947. PMID 21445376
- [Result] Laperriere A, Ironson GH, Antoni MH, Pomm H, Jones D, Ishii M, Lydston D, Lawrence P, Grossman A, Brondolo E, Cassells A, Tobin JN, Schneiderman N, Weiss SM. Decreased depression up to one year following CBSM+ intervention in depressed women with AIDS: the smart/EST women's project. J Health Psychol. 2005 Mar;10(2):223-31. doi: 10.1177/1359105305049772. PMID 15723892
- [Result] Ironson G, Weiss S, Lydston D, Ishii M, Jones D, Asthana D, Tobin J, Lechner S, Laperriere A, Schneiderman N, Antoni M. The impact of improved self-efficacy on HIV viral load and distress in culturally diverse women living with AIDS: the SMART/EST Women's Project. AIDS Care. 2005 Feb;17(2):222-36. doi: 10.1080/09540120512331326365. PMID 15763716
- [Result] Segal-Isaacson CJ, Tobin JN, Weiss SM, Brondolo E, Vaughn A, Wang C, Camille J, Gousse Y, Ishii M, Jones D, Laperriere A, Lydston D, Schneiderman N, Ironson G. Improving dietary habits in disadvantaged women with HIV/AIDS: the SMART/EST women's project. AIDS Behav. 2006 Nov;10(6):659-70. doi: 10.1007/s10461-006-9115-5. Epub 2006 Jun 1. PMID 16770694
- [Result] Weiss SM, Tobin JN, Lopez M, Simons H, Cook R, Jones DL. Translating an Evidence-Based Behavioral Intervention for Women Living with HIV into Clinical Practice: The SMART/EST Women's Program. Int J Behav Med. 2015 Jun;22(3):415-24. doi: 10.1007/s12529-014-9399-1. PMID 24623475
- [Result] Jones DL, Lopez M, Simons H, Diaz-Gloster M, Tobin JN, Weiss SM. Translation of a comprehensive health behavior intervention for women living with HIV: the SMART/EST Women's Program. Transl Behav Med. 2013 Dec;3(4):416-25. doi: 10.1007/s13142-013-0213-4. PMID 24294330
- [Result] Webel AR. Testing a peer-based symptom management intervention for women living with HIV/AIDS. AIDS Care. 2010 Sep;22(9):1029-40. doi: 10.1080/09540120903214389. PMID 20146111
- See also: Clinical Directors Network website for previous iterations of the SMART/EST group for HIV-positive women — https://www.cdnetwork.org/smart-est